CLINICAL TRIAL: NCT03456284
Title: Pilot Study to Assess Safety and Feasibility of Normothermic Machine Perfusion to Preserve and Evaluate Orphan Livers
Brief Title: Safety and Feasibility of Normothermic Machine Perfusion to Preserve and Evaluate Orphan Livers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Koji Hashimoto, Staff Physician, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Orphan liver
Record Dates: First submitted 2018-02-15; First posted 2018-03-07 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Normothermic Liver perfusion (Experimental): This group has the liver grafts preserved using the Normothermic Liver perfusion Device
  Interventions: Device: Normothermic Liver perfusion

INTERVENTIONS:
Device: Normothermic Liver perfusion — The liver grafts will be preserved and evaluated at physiological temperature and have continuous perfusion with oxygen and nutrient supply in the ex vivo organ preservation phase

SUMMARY:
Orphan livers are organs that have been declined for clinical use by all centers due to their marginality. The current standard of care of liver preservation before transplant is cold storage. NMP may allow these livers to be evaluated before transplantation. NMP has already been used in a clinical setting with promising results. The advantage to utilizing NMP is that it would attenuate the incidence and clinical impact of classical preservation injury, allow liver function assessment before implantation and thus improve donor pool and outcomes for high risk ECD liver transplants performed at our center.

DETAILED DESCRIPTION:
This will be a single center prospective cohort pilot study. 30 livers that have been declined for clinical use by all centers due to their marginality will be preserved with NMP in 1-18 hours after cross clamp and cold flush. The liver grafts at NMP will be at Physiological temperature and have oxygen and nutrient supply with continuous perfusion. Once the liver grafts have been evaluated and determined to be transplantable, the transplantation and post-transplant care will follow the standard of care. The follow-up period is 12 months after transplantation. The primary end point will be the rate of patient survival and primary non function (PNF) within 30 days after transplantation, while the secondary end points will be: Early Allograft Dysfunction (EAD), 6 months patient and graft survival, peak liver function tests in the first 7 days after transplantation, surgical outcomes (operative time, transfusion requirement etc.), rate of post-transplant kidney failure, assessment of histological ischemia reperfusion (liver and bile duct), rate of vascular complications, rate of biliary complications, hospital and ICU length of stay, rejection rate, infection rate, the ability to predict function based on "on-pump" viability markers, and the incidence of adverse effect (AE).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary liver transplantation
* Age 18-75 years at the time of transplantation
* Willingness and ability to comply with the study procedures
* Signed Informed Consent Form
* For patients with hepatocellular carcinoma as indication for Orthoptic Liver Transplantation (OLT), tumor must be within Milan Criteria or down-staged to Milan Criteria.

Exclusion Criteria:

Recipient Exclusion Criteria:

* History of prior solid organ transplantation
* Patient on a respiratory and/or cardiocirculatory support at the time of transplant
* MELD score >35
* HIV positive patient
* Patient with current severe systemic infection
* Multiorgan transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The rate of patient survival | 30 days post-transplantation
The rate of primary non-function | 30 days post-transplantation
  primary non-function is defined as non life sustaining liver function requiring retransplantation or leading to death with 30 days after transplantation

SECONDARY OUTCOMES:
The rate of Early Allograft Dysfunction post-transplantation | 7 days post-transplantation
  The presence of at least one of the following at post-transplant 7 days: serum bilirubin >= 10 mg/dL, international normalized ratio (INF) >= 1.6; and/or aspartate aminotransferase (AST) > 2000 U/L at any time in the first 7 posttransplant days (POD)
graft survival | 6 months post-transplantation
  The allograft will be considered lost if a patient has a liver re-transplant or in the event of patient death.
peak aspartate aminotransferase (AST) in the first 7 days post-transplantation | in the first 7 days post-transplantation
  CLINICAL LABORATORY TEST
peak Alanine Aminotransferase (ALT) in the first 7 days post-transplantation | in the first 7 days post-transplantation
  CLINICAL LABORATORY TEST
peak bilirubin in the first 7 days post-transplantation | in the first 7 days post-transplantation
  CLINICAL LABORATORY TEST

CONTACTS AND LOCATIONS:
Overall Officials: Koji Hashimoto, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No